CLINICAL TRIAL: NCT01809678
Title: Efficacy of Yoga as a Complementary Therapy for Smoking Cessation
Brief Title: Yoga as a Complementary Therapy for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Beth Bock, Ph.D., Staff Psychologist, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AT006948 (NIH)
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Tobacco Dependence
Keywords: Smoking; Tobacco; Yoga
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Yoga; Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Smoking Cessation plus Yoga (Experimental): Twice weekly, 1-hour yoga classes delivered for 8 weeks combined with once-weekly, 1-hour cognitive-behavioral smoking cessation classes.
  Interventions: Behavioral: Smoking Cessation; Behavioral: Yoga
- Smoking Cessation plus Wellness (Active Comparator): Twice-weekly, 1-hour Wellness classes given on a variety of health topics twice weekly to match schedule of the yoga classes, plus 1-hour per week of cognitive-behavioral smoking cessation
  Interventions: Behavioral: Smoking Cessation; Other: Wellness

INTERVENTIONS:
Behavioral: Smoking Cessation — Once weekly program of cognitive-behavioral therapy for smoking cessation
Behavioral: Yoga — Twice weekly program of 1-hour Iyengar yoga classes
  Arms: Smoking Cessation plus Yoga
Other: Wellness — Twice weekly program of 1-hour wellness classes on a variety of health topics.
  Arms: Smoking Cessation plus Wellness

SUMMARY:
This study examines the efficacy of yoga as a complementary therapy for smoking cessation

DETAILED DESCRIPTION:
Despite the existence of effective medications for smoking cessation, approximately 50-80% of smokers attempt to quit without using pharmacotherapy. Efforts to encourage medication use during cessation attempts have met with mixed success. Many do not use medications because of concerns about side effects, contraindications that make medication use inappropriate, and individual preferences for chemical-free quit attempts. This leaves many smokers seeking an effective alternative to assist them in attempting to quit smoking. Each year, over 41% of smokers report failed attempts to quit smoking. Thus, effective non-pharmacological interventions to increase rates of successful cessation are greatly needed.

Our research, and the research of other investigators, has demonstrated that traditional (Western) exercise (e.g., brisk walking, bicycling) improves smokers' ability to successfully quit. Exercise may help smokers quit by reducing concerns regarding post-cessation weight gain, and by reducing nicotine withdrawal and enhancing mood. Recent research suggests that yoga is an acceptable and potentially effective alternative therapy for smoking cessation for several reasons: As a form of exercise, yoga shares many of the same properties as traditional (Western) aerobic exercise in that yoga has been shown to improve mood, physical fitness, weight control, self-image and quality of life in healthy and ill populations. Moreover, features of yoga, including a focus on breathing, mental concentration, meditation, stress reduction and enhanced mood are likely to have special relevance for smokers who are trying to quit. Thus, yoga may be particularly attractive as an alternative for individuals who either cannot use medications, or who choose not to use medications while quitting.

The proposed study will test the efficacy of Yoga as a complementary therapy for smoking cessation using a randomized, controlled study design. Adult smokers will be randomly assigned to either; 1) Yoga, or 2) an equal contact time Control group (CTL) given a health & wellness program to control for contact time. All participants will be provided (separately by treatment group assignment) with the same cognitive-behavioral Smoking Cessation Counseling (SCC). Smoking abstinence will be measured at the end of treatment (week 8) and at 3, 6 and 12 months follow-up. We hypothesize that abstinence will be significantly higher in the SCC+Yoga group compared to SCC+CTL. We will also test theoretically posited mediators of intervention efficacy (e.g., perceived stress, cognitive/perceptual changes), examine the cost-efficacy of the yoga intervention, and examine the relationship between maintenance of yoga practice during the post-treatment period and smoking status. This study builds on our programmatic line of research developing innovative, theory-driven smoking cessation therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older (physician clearance for age > 65)
* English-speaking
* Currently Healthy
* Smoking smoked 5 or more cigarettes/day
* Must accept randomization procedure
* BMI< 40
* Will be Living in RI/MA/CT for next year

Exclusion Criteria:

* Participated in any Yoga, Tai Chi, Qi Gong or Mindfulness-based therapy program twice in the past month or 10 times within the past year
* MD refused consent or Unable to obtain MD consent
* Unable to attend program due to work or home schedule
* Currently using medications or in active treatment to quit smoking
* Currently or planned participation in research or treatment programs that would interfere with this study
* Presence of health conditions that would make participation in yoga difficult or dangerous

Medical Exclusion Criteria

* Cardiovascular disease
* Stroke/TIA
* Chest pain with physical activity
* Current or recent (< 6 months) cancer treatment
* Uncontrolled Hypertension
* Untreated major depression or hospitalization < six months
* Bone joint problems
* Liver or Kidney Disease
* Fainting within the past year
* History of seizures
* Balance condition that interferes with ability to exercise
* Respiratory Condition - COPD (e.g., emphysema requiring oxygen)
* Liver Disease
* Kidney Disease
* Other medical condition that would interfere with ability to exercise
* Hypothyroid (not on stable medication for 3 months)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence | One year
  Abstinence from smoking at 1-year post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Background] Thind H, Jennings E, Fava JL, Sillice MA, Becker BM, Hartman SJ, Bock BC. Differences between Men and Women Enrolling in Smoking Cessation Programs Using Yoga as a Complementary Therapy. J Yoga Phys Ther. 2016;6(3):245. doi: 10.4172/2157-7595.1000245. Epub 2016 Jun 15. PMID 27683623
- [Background] Bock BC, Rosen RK, Fava JL, Gaskins RB, Jennings E, Thind H, Carmody J, Dunsiger SI, Gidron N, Becker BM, Marcus BH. Testing the efficacy of yoga as a complementary therapy for smoking cessation: design and methods of the BreathEasy trial. Contemp Clin Trials. 2014 Jul;38(2):321-32. doi: 10.1016/j.cct.2014.06.003. Epub 2014 Jun 14. PMID 24937018
- [Result] Bock BC, Dunsiger SI, Rosen RK, Thind H, Jennings E, Fava JL, Becker BM, Carmody J, Marcus BH. Yoga as a Complementary Therapy for Smoking Cessation: Results From BreathEasy, a Randomized Clinical Trial. Nicotine Tob Res. 2019 Oct 26;21(11):1517-1523. doi: 10.1093/ntr/nty212. PMID 30295912
- [Result] Bock BC, Thind H, Dunsiger S, Fava JL, Jennings E, Becker BM, Marcus BH, Rosen RK, Sillice MA. Who Enrolls in a Quit Smoking Program with Yoga Therapy? Am J Health Behav. 2017 Nov 1;41(6):740-749. doi: 10.5993/AJHB.41.6.8. PMID 29025502
- [Result] Rosen RK, Thind H, Jennings E, Guthrie KM, Williams DM, Bock BC. "Smoking Does Not Go With Yoga:" A Qualitative Study of Women's Phenomenological Perceptions During Yoga and Smoking Cessation. Int J Yoga Therap. 2016 Jan;26(1):33-41. doi: 10.17761/1531-2054-26.1.33. PMID 27797659